CLINICAL TRIAL: NCT03969797
Title: Quality Feedback of 19 Cases by AED Operation in Out-of-hospital Environment: a Prospective Randomized Log Analysis
Brief Title: AED Log Analysis of 19 Cases in Out-of-hospital Environment
Status: Completed | Type: Observational
Sponsor: RadianQbio (Industry)
Responsible Party: Sponsor
Other Study IDs: HR501_20190527
Record Dates: First submitted 2019-05-27; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Arrest, Sudden
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 32 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RADIAQBIO Heart Guardian HR-501 — Arm one offers ECG data and electric shocks recorded during AED operation.

SUMMARY:
The study performed to demonstrate a reasonable assurance of safety and effectiveness of the Heart Guardian HR-501 when used in an out-of-hospital environment.

DETAILED DESCRIPTION:
The defibrillation study was conducted by analyzing the logs of Heart Guardian HR-501 with Radian ECG Viewer. The product analysis was studied whether the device was operated normally in ECG analysis and electric shocks.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest
* > 12 months

Exclusion Criteria:

* age under 12 months

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients using AED HR-501
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Identification ECG from patients | during operating, approximately 2 hours
  The AED identifies if ECG is VF or normal

SECONDARY OUTCOMES:
Survival patients by electric shock | 24 hours
  Ratio of patients were survived after electric shock delivered

CONTACTS AND LOCATIONS:
Locations (1):
- Radianqbio, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No